CLINICAL TRIAL: NCT05997082
Title: Mindful Self-compassion, Compassion Fatigue, Secondary Traumatic Stress, and Burnout Among Specialist Rehabilitation Providers - a Mixed Methods Study Protocol
Brief Title: A Mindful Self-compassion Based Intervention for Specialist Rehabilitation Providers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Robert Simpson, Physiatrist and Associate Scientist, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 5492
Record Dates: First submitted 2023-08-10; First posted 2023-08-18 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Burnout, Professional; Compassion Fatigue; Secondary Traumatic Stress
Keywords: Mindful Self-Compassion; Compassion-Based Intervention; Meditation; Online Intervention; Rehabilitation Providers; Physiatrists
MeSH Terms: conditions — Burnout, Professional; Compassion Fatigue

STUDY DESIGN:
Masking Description: No masking since there is only 1 group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Participants in the intervention (Experimental): Participants in the intervention will participate in the 6-week mindfulness self-compassion course delivered online.
  Interventions: Other: Mindfulness Self-Compassion Course

INTERVENTIONS:
Other: Mindfulness Self-Compassion Course — This course is designed to reduce burnout and compassion fatigue among specialist rehabilitation providers. Course materials are adapted from the Center for Mindful Self-Compassion (CMSC).

SUMMARY:
The goal of this clinical trial is to explore the impact of an online compassion-based intervention on burnout among specialist rehabilitation providers. Post-intervention interviews aim to gather information on: burnout and compassion, experiences with the intervention, barriers and facilitators to taking part, and suggestions for improving online course delivery.

DETAILED DESCRIPTION:
Burnout threatens the sustainability of compassionate care in rehabilitation. This project explores the impact of an online compassion-based intervention on burnout among specialist inpatient rehabilitation healthcare providers. Thirty specialist rehabilitation healthcare providers will be recruited to take part. The online intervention will include six weekly live one-hour sessions. Healthcare provider socio-demographic, practice, and wellness measures will be collected at baseline, post-course, and three months later. Qualitative interviews will be used to explore participant views on burnout and compassion, experiences with the intervention, barriers and facilitators to taking part, and suggestions for improving online course delivery. Up to two instructors and support persons will be invited to participate in qualitative interviews to explore their views for improving online course delivery.

ELIGIBILITY:
Inclusion Criteria:

* Employed substantively as a regulated health professional (e.g., physiatrist, nurse, allied health professional) by a specialist rehabilitation institute (e.g., Sunnybrook/St. John's Rehab, University Hospital Network, Providence Healthcare, Westpark Healthcare)
* Over 18 years of age
* Able to speak, read, and write in English
* Willing to take part in the MSC course for up to the full 6-week duration
* Willing to complete all study related questionnaires

Exclusion Criteria:

* Those already having completed a MSC (mindfulness-based stress reduction) course or mindfulness-based cognitive therapy within the past 12 months
* Those employed as agency staff

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2023-08-17 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Professional Quality of Life Scale (ProQOL) Version 5 | Baseline, post-intervention (6 weeks after baseline), and 3 months post-intervention
  Measures the positive and negative effects of one's compassion for those that they help rehabilitate.

SECONDARY OUTCOMES:
Relational Compassion Scale | Baseline, post-intervention (6 weeks after baseline), and 3 months post-intervention
  Measure's ones tendencies for receiving and providing relational compassion.
Self-Compassion Scale - Short Form | Baseline, post-intervention (6 weeks after baseline), and 3 months post-intervention
  Measures how one typically acts towards themselves in difficult times.
The Brief Interpersonal Reactivity Index | Baseline, post-intervention (6 weeks after baseline), and 3 months post-intervention.
  Measures the different ways that people may think about their lives.
5 Facet Mindfulness Questionnaire: Short Form | Baseline, post-intervention (6 weeks after baseline), and 3 months post-intervention
  Measures one's tendencies to engage in mindfulness practices.
Perceived Stress Scale | Baseline, post-intervention (6 weeks after baseline), and 3 months post-intervention
  Measures one's thoughts and feelings pertaining to stress.
Difficulties in Emotion Regulation Scale - Short Form | Baseline, post-intervention (6 weeks after baseline), and 3 months post-intervention
  Measures emotion regulation.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Simpson, Md, PhD, Principal Investigator — Sunnybrook Research Institute
Locations (1):
- St. John's Rehab (Sunnybrook Health Sciences Centre), Toronto, Ontario, Canada